CLINICAL TRIAL: NCT05022459
Title: Prevention of Bleeding in Patients With Moderate and Severe Hemophilia A Playing Sports: A Comparison Between Factor VIII and Emicizumab Prophylaxis -STEP: SporTs Emicizumab Prophylaxis
Brief Title: Prevention of Bleeding in Patients With Moderate and Severe Hemophilia A Playing Sports: A Comparison Between Factor VIII and Emicizumab Prophylaxis
Acronym: STEP
Status: Recruiting | Type: Observational
Sponsor: Wayne State University (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Principal Investigator, Meera Chitlur, Director, Hemophilia Treatment Center and Hemostasis Program, Principal Investigator, Clinical Professor, Wayne State University
Other Study IDs: STEP Study
Record Dates: First submitted 2021-08-23; First posted 2021-08-26 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Hemophilia A
MeSH Terms: conditions — Hemophilia A | interventions — emicizumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Participants will have the option to agree to allow any blood leftover from study testing to be stored for future research.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (2):
- Emicizumab Prophylaxis: This group will include patients on standard of care Emicizumab prophylaxis for Hemophilia A
  Interventions: Drug: Emicizumab
- FVIII Prophylaxis: This group will include patients on standard of care FVIII prophylaxis for Hemophilia A
  Interventions: Drug: FVIII

INTERVENTIONS:
Drug: Emicizumab — Patients in this group will be on standard of care Emicizumab prophylaxis for Hemophilia A
  Groups: Emicizumab Prophylaxis
Drug: FVIII — Patients in this group will be on standard of care FVIII prophylaxis for Hemophilia A
  Groups: FVIII Prophylaxis

SUMMARY:
Hemophilia A (HA) is a genetic bleeding disorder resulting from a deficiency or absence of factor VIII (FVIII), which is necessary in the clotting process. This disorder occurs mostly in males and in severe cases causes frequent bleeding episodes in joints and muscles which can lead to progressive damage that affects mobility and quality of life. Prophylactic FVIII administered intravenously every other day has been the standard of care treatment for HA for the past few decades.

Sports and physical activity are generally encouraged in patients with hemophilia on appropriate prophylactic treatment to increase strength, prevent or decrease obesity, accrue and maintain bone density and encourage normal socialization. To ensure safety with participation in sports in persons with hemophilia A (PWHA), timing of FVIII administration is often adjusted to maximize FVIII at the time of sports. The exact factor level that is needed to safely participate in sports and minimize bleeding risk is not yet known. Based on clinical practice, infusion of FVIII to near the lower limit of normal right before participation in sports generally works to prevent bleeding.

The study is looking at how well the newly approved medication Emicizumab works compared to Factor VIII to prevent bleeding in patients with Hemophilia A who play sports. The study will enroll children and adolescents who are already on Emicizumab or Factor VIII who are currently playing sports.

DETAILED DESCRIPTION:
Hemophilia A (HA) is a genetic bleeding disorder resulting from a deficiency or absence of factor VIII (FVIII) which is necessary in the clotting process. This disorder occurs mostly in males and in severe cases causes frequent bleeding episodes in joints and muscles which can lead to progressive damage that affects mobility and quality of life. Intravenous prophylactic (preventative) treatment is the standard of care used in minimizing bleeding events and complications. Since the 1990s recombinant FVIII (rFVIII) concentrates have been standard of care treatment options for patients with hemophilia A. Prophylactic treatment is burdensome because it requires self-administered intravenous infusions several (3-4) times a week and prophylactic FVIII does not completely prevent bleeding.

Sports and physical activity are generally encouraged in patients with hemophilia on appropriate prophylactic treatment to increase strength, prevent or decrease obesity, accrue and maintain bone density and encourage normal socialization. To ensure safety with participation in sports in persons with hemophilia A (PWHA), timing of FVIII administration is frequently adjusted to maximize FVIII at the time of sports. The exact factor level that is needed to safely participate in sports and minimize bleeding risk is not yet known. Based on clinical practice, infusion of FVIII to near the lower limit of normal right before participation in sports generally works to prevent bleeding.

Emicizumab is an engineered antibody that mimics what activated factor VIII does in the blood to help it clot. Emicizumab is an antibody and is present in the blood for a long time and approximately 50% of an injected dose is still circulating in the blood 4 weeks later; this permits less frequent dosing (Anywhere from once a week to once every 4 weeks). Emicizumab can be injected under the skin (subcutaneous) instead of having to be injected into a vein (intravenous). Emicizumab's convenience compared to FVIII, reduced bleeding rate, and in many cases decreased annual cost, have led to its adoption by many patients with HA. Emicizumab does not completely normalize hemostasis (the physiological process that stops bleeding) and although the exact comparison of hemostatic correction on maintenance doses of Emicizumab to that with FVIII replacement cannot be determined with existing assays, it has been clinically demonstrated that Emicizumab changes the bleeding characteristics of a patient with severe hemophilia A to a milder profile. While this may provide sufficient protection to prevent spontaneous bleeding into the joints, it remains unknown if this is sufficient to prevent activity/sports related joint bleeds (especially activities with moderate to high risk of bleeding).

A disadvantage of Emicizumab prophylaxis is that the steady state produced with Emicizumab prophylaxis does not allow dosing at the time of sports participation. One major question is whether the "steady state" levels of hemostasis achieved with Emicizumab are enough to prevent joint damage with sports participation, and whether there is a threshold of participant age or size or activity intensity above which Emicizumab is not generally adequate.

Emicizumab use permits maintenance of "steady state" hemostasis in the range of mild hemophilia without frequent infusions. Studying patients taking Emicizumab while engaging in sports permits us to study the effects of participation in physical activity with steady state hemostasis levels in the range of mild hemophilia compared to peak hemostatic levels from factor infusions given immediately before engaging in activity/sports. This is a crucial factor in the decision-making process for physicians making treatment recommendations to optimize preventive therapy for physically active people with hemophilia A.

The purpose of this investigator-initiated study is to better understand the safety of sports in people with Hemophilia A, the breakthrough bleed rates, and the types of bleeds related to sports activities in patients on Emicizumab vs traditional FVIII prophylaxis. This information will help in the decision-making process for physicians making treatment recommendations for physically active people with hemophilia A.

ELIGIBILITY:
Inclusion Criteria:

1. Participant (if 18 years of age or older) or parent/LAR is willing and able to provide written informed consent; minor participant is willing and able to provide assent, if applicable based on site and local regulations
2. Males and females between 6 to ≤ 19 years of age at time of enrollment with moderate to severe Hemophilia A (FVIII activity ≤ 5%) without inhibitors are eligible for participation in this study
3. Participants must be on Emicizumab or standard FVIII prophylaxis per institutional/primary hematologist recommendations
4. Participants must be engaging in or registered to start participating in one or more sports activities with moderate to high risk of bleeding as defined by the NHF- Playing it Safe guidelines (numerical rating >/= 2).
5. Participant must be willing to keep activity, bleed, and treatment logs for the duration of the study

Exclusion Criteria:

1. Participant/parent/LAR unwilling to provide informed consent/assent
2. Unwilling to log or document bleeds and treatment information as per study guidelines
3. Participants with any other bleeding disorders will be excluded
4. Patients who are pregnant, planning to become pregnant, or breastfeeding should not be enrolled in the study
5. Participants on concomittent FVIII replacement and emicizumab for sports participation

Ages: 6 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: This study will enroll patients who are already on Emicizumab or FVIII prophylaxis as per standard of care and who are already participating in sports activities with moderate to high risk of bleeding.
Sampling Method: Non-Probability Sample
Enrollment: 72 (Estimated)
Dates: Start 2023-08-16 (Actual); Primary Completion 2029-01 (Estimated); Study Completion 2029-03 (Estimated)

PRIMARY OUTCOMES:
Number of bleeds | 2 years
  Number of bleeds without trauma, during participation in sports activities

SECONDARY OUTCOMES:
Change in HJHS scores | 3 years
  Change in Hemophilia Joint Health Scores (HJHS). The HJHS provides a total score (higher score is worse; max=124), joint specific scores, and a global gait score.
Change in bone mineral density | 3 years
  Change in bone mineral density as measured by DEXA Scan
Change in biomarkers of bone and joint health | 3 years
  Change in biomarkers of bone and joint health as measured by (sRANKL (osteoclastogenesis), CTX-1 (Bone resorption), CS846 (cartilage repair) and IL-1 beta, IL6 and TNF-alpha (markers of inflammation).
Number of FVIII doses for breakthrough bleeding episodes | 3 years
  Number of doses of factor needed to treat breakthrough bleeding episodes
MRI changes in relevant joints | 3 years
  MRI changes in relevant joints (The joint to be imaged will be determined based on the sport activity; joints most involved in the activity will be imaged).

CONTACTS AND LOCATIONS:
Overall Officials: Meera Chitlur, MD, Principal Investigator — Wayne State University
Locations (9):
- United States (9):
  - Arkansas Children's Hospital, Little Rock, Arkansas
  - Stanford University, Palo Alto, California
  - Rady Children's Hospital, San Diego, California
  - Johns Hopkins All Children's Hospital, St. Petersburg, Florida
  - Indiana Hemophilia & Thrombosis Center, Indianapolis, Indiana
  - Boston Children's Hospital, Boston, Massachusetts
  - Children's Hospital of Michigan, Detroit, Michigan
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Oklahoma Center for Bleeding and Clotting Disorders, Oklahoma City, Oklahoma

IPD SHARING:
Plan to Share IPD: No